



## MERINO:2 | EN EKSTRA OPPFØLGING AV DELTAKERE I MERINO-STUDIEN

#### FORMÅLET MED PROSJEKTET OG HVORFOR DU BLIR SPURT

Dette er et spørsmål til deg om å delta i en oppfølgingsundersøkelse etter MERINO-studien på Diakonhjemmet sykehus. Vi ønsker å ta et <u>røntgenbilde av hendene dine</u> samt at du hjemme besvarer <u>noen spørreskjemaer</u> <u>om symptomer fra din artrose</u>.

Hensikten er å sammenlikne langtidseffektene av legemiddelet metotreksat med behandling som vanlig. Det er ingen andre studier som undersøker langtidseffektene av metotreksat. Derfor inviterer vi alle deltakere fra MERINO-studien til en ekstra oppfølging 2,5 år etter man ble med i MERINO. Vi vil sammenlikne med den første datainnsamling fra MERINO-studien, og derfor går denne forespørselen <u>til alle som ble rekruttert i MERINO-studien</u>, uavhengig om de fullførte eller ikke.

Studien utgår fra revmatologisk avdeling på Diakonhjemmet sykehus og ledes av Alexander Mathiessen.

Status på den opprinnelige MERINO-studien: Per oktober 2024 er 131 av 153 deltakere i MERINO-studien rekruttert og vi håper å komme i mål i løpet av februar 2025. Vi planlegger nå hovedanalysen som gjøres når alle rekrutterte deltakere har nådd 6 måneders behandling.

## HVA INNEBÆRER PROSJEKTET FOR DEG?

Dersom du sier deg villig til å være med i studien vil du 1) kalles inn til et røntgenbilde av hendene dine ca 2,5 år etter du ble rekruttert til MERINO-studien og 2) få en lenke for besvarelse av noen spørreskjemaer i Nettskjema. Disse kan du fylle ut hjemme på mobil eller pc og krever sikker innlogging med BankID. Vi vil sammenlikne med data fra den opprinnelige studien, samt innhente informasjon om hvilke legemidler deltagerne har brukt i denne periode fra Legemiddelregisteret.

### MULIGE FORDELER OG ULEMPER

MERINO:2 innebærer bruk av din tid, i form av et oppmøte for røntgenbilde og besvarelse av spørreseskjemaer. For de som bor i nærheten av Oslo vil røntgenbilde bli tatt på Diakonhjemmet sykehus, mens de som bor lenger unna vil få innkallelse til et røntgeninstitutt nær eget bosted.

- Røntgen av hender tilsvarer minimalt med stråling, ca. 3 timer med naturlig bakgrunnsbestråling som vi utsettes for daglig.
- Spørreskjemaene er begrenset til å ta omtrent 15 minutter.

Vi ser ingen direkte fordeler for deg som individ ved disse undersøkelsene, men på gruppenivå gir dette verdifulle supplerende data.

# FRIVILLIG DELTAKELSE OG MULIGHET FOR Å TREKKE DITT SAMTYKKE

Det er frivillig å delta i prosjektet. Dersom du ønsker å delta, undertegner du samtykkeerklæringen. Du kan når som helst og uten å oppgi noen grunn trekke ditt samtykke. Det vil ikke ha noen negative konsekvenser for deg eller din behandling hvis du ikke vil delta eller senere velger å trekke deg. Dersom du trekker tilbake

samtykket, vil det ikke forskes videre på dine opplysninger. Du kan kreve innsyn i opplysningene som er lagret om deg, og disse vil da utleveres innen 30 dager. Du kan også kreve at dine opplysninger i prosjektet slettes.

Adgangen til å kreve sletting eller utlevering gjelder ikke dersom opplysningene er anonymisert eller publisert. Denne adgangen kan også begrenses dersom opplysningene er inngått i utførte analyser.

Dersom du senere ønsker å trekke deg eller har spørsmål til prosjektet, kan du kontakte prosjektleder (se kontaktinformasjon på siste side).

#### HVA SKJER MED OPPLYSNINGENE OM DEG?

Opplysningene som registreres om deg skal kun brukes slik som beskrevet under formålet med prosjektet. Etter at forskningsprosjektet er ferdig, vil opplysningene om deg bli oppbevart i fem år av kontrollhensyn. Eventuelle utvidelser i bruk og oppbevaringstid kan kun skje etter godkjenning fra regionale komiteer for medisinsk og helsefaglig forskningsetikk (REK) og andre relevante myndigheter.

Du har rett til innsyn i hvilke opplysninger som er registrert om deg og rett til å få korrigert eventuelle feil i de opplysningene som er registrert. Du har også rett til å få innsyn i sikkerhetstiltakene ved behandling av opplysningene. Du kan klage på behandlingen av dine opplysninger til Datatilsynet og institusjonen sitt personvernombud.

Alle opplysningene vil bli behandlet uten navn og fødselsnummer eller andre direkte gjenkjennende opplysninger (=kodede opplysninger). En kode knytter deg til dine opplysninger gjennom en navneliste. Listen som kan koble ditt navn til koden vil kun bli oppbevart på Diakonhjemmet sykehus og bare personell som har ansvar for studien har tilgang til denne listen.

Publisering av resultater er en nødvendig del av forskningsprosessen og gjøres på sammenstilte data slik at man som individ ikke kan bli gjenkjent.

#### DELING AV OPPLYSNINGER OG OVERFØRING TIL UTLANDET

Som en del av gjennomføringen av studien kan det bli aktuelt å overføre innsamlede opplysninger til internasjonale samarbeidspartnere i dette prosjektet, både innenfor EU/EØS og utenfor EU/EØS (Storbritannia og USA). I slike tilfeller vil dataene være avidentifiserte (spørreskjemaer og røntgen-bilder), hvor formålet er å gjøre analyser av forskningsspørsmål som er beskrevet i dette samtykkeskjemaet. Diakonhjemmet sykehus er ansvarlig for at overføringen av opplysninger skjer i samsvar med norsk rett og EU sin personvernlovgivning (GDPR). Koden som knytter deg til dine personidentifiserbare opplysninger vil ikke bli utlevert. Informasjon om slikt internasjonalt samarbeid og overføring skal være tilgjengelig når det skjer, løpende informasjon kan finnes her: www.remedy-senter.no/project/merino.

# FORSIKRING

Du er forsikret i henhold til Norsk Pasientskadeerstatning (pasientskadeloven).

### **ØKONOMI**

Det påløper ikke kostnader for deg å delta i studien. Alle utgifter dekkes av sponsor Diakonhjemmet Sykehus. Eventuelle reiseutgifter vil dekkes.

## GODKJENNINGER

Regional komité for medisinsk og helsefaglig forskningsetikk (REK) har gjort en forskningsetisk vurdering og godkjent prosjektet (REK 2024/715758).

Etter ny personopplysningslov har behandlingsansvarlig for dine personopplysninger Diakonhjemmet Sykehus og prosjektleder Alexander Mathiessen et selvstendig ansvar for å sikre at behandlingen av dine opplysninger

har et lovlig grunnlag. Dette prosjektet har rettslig grunnlag i EUs personvernforordning artikkel 6 a og 9 nr. 2 a og ditt samtykke. Du har rett til å klage på behandlingen av dine opplysninger til Datatilsynet.

## KONTAKTOPPLYSNINGER

Dersom du har spørsmål til prosjektet, opplever uønskede hendelser eller bivirkninger, eller ønsker å trekke deg fra deltakelse, kan du kontakte prosjektleder Alexander Mathiessen:

Telefon 97501889

Mail <u>a-mathi1@diakonsyk.no</u>

Dersom du har spørsmål om personvernet i prosjektet, kan du kontakte personvernombudet ved institusjonen: <a href="mailto:personvern@diakonsyk.no">personvern@diakonsyk.no</a>.

JEG SAMTYKKER TIL Å DELTA I PROSJEKTET OG TIL AT MINE PERSONOPPLYSNINGER BRUKES SLIK DET ER BESKREVET

| Sted og dato | Deltakers signatur |
|--------------|-------------------------------------|
| | Deltakers navn med trykte bokstaver |